CLINICAL TRIAL: NCT06800521
Title: Mixed Reality as a Health Literacy Strategy for Breastfeeding Education: A Randomized Controlled Trial
Brief Title: Mixed Reality as a Health Literacy Strategy for Breastfeeding Education
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad de la Sabana (Other)
Responsible Party: Principal Investigator, sergio Ivan agudelo Perez, Assistant Professor, Universidad de la Sabana
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: MEDESP-27-2024
Record Dates: First submitted 2025-01-15; First posted 2025-01-30 (Actual); Last update posted 2025-01-30 (Actual); Status verified 2025-01

CONDITIONS: Breastfeeding Education; Maternal Self-Efficacy; Breastfeeding Satisfaction
Keywords: Breastfeeding; Health Education; Self-Efficacy; Maternal-Child Health
MeSH Terms: conditions — Breast Feeding; Health Education

STUDY DESIGN:
Intervention Model Description: This study uses a parallel assignment model, where participants are randomly assigned to one of two groups: the intervention group receiving a mixed reality-based educational strategy or the control group receiving traditional breastfeeding counseling. Both groups will be followed independently throughout the study period to evaluate and compare outcomes, including breastfeeding satisfaction, self-efficacy, and adherence to exclusive breastfeeding during the first week postpartum. Randomization will ensure comparable baseline characteristics between groups, and the study design allows for the direct evaluation of the intervention's effectiveness.
Who Masked: Investigator
Masking Description: Due to the nature of the intervention, participants could not be masked to their group assignment. However, the investigators responsible for analyzing the data were masked to the group allocations. This approach ensures that the statistical analysis and interpretation of results remain unbiased, despite the lack of masking at the participant level.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Mixed Reality Educational Intervention (Experimental): Participants in this arm will receive a mixed reality-based educational intervention, including:
  Mixed Reality Goggles: Simulating breastfeeding scenarios. Immersive Audio-Visual Materials: Enhancing engagement and understanding. Realistic Breastfeeding Simulations: Providing hands-on practice to build confidence.
  Delivered in a single session during the third trimester, this intervention aims to improve breastfeeding satisfaction and self-efficacy.
  Follow-Up:
  Satisfaction and self-efficacy will be assessed using MBFES and BSES-SF. Exclusive breastfeeding adherence will be monitored during the first postpartum week.
  Interventions: Behavioral: Mixed Reality Breastfeeding Education
- Traditional Breastfeeding Counseling (Active Comparator): Participants in this arm will receive traditional breastfeeding counseling as part of routine prenatal care. The session includes verbal and visual education by trained healthcare professionals, focusing on breastfeeding techniques, benefits, and solutions to common challenges.
  Delivered during the third trimester, this approach represents the standard of care.
  Follow-Up: Breastfeeding satisfaction and self-efficacy will be assessed using MBFES and BSES-SF.
  Adherence to exclusive breastfeeding will be monitored during the first postpartum week.
  Interventions: Behavioral: Traditional Breastfeeding Counseling

INTERVENTIONS:
Behavioral: Mixed Reality Breastfeeding Education — Mixed Reality Breastfeeding Education:
  This intervention includes an innovative mixed reality-based educational strategy combined with traditional breastfeeding counseling. Participants use mixed reality goggles to experience immersive breastfeeding scenarios, interact with audio-visual materials tailored for breastfeeding education, and engage with realistic breastfeeding simulations. The session is delivered once during the third trimester of pregnancy and lasts approximately 90 minutes. This intervention is designed to improve maternal confidence, satisfaction, and adherence to exclusive breastfeeding through an engaging and practical learning environment.
  Arms: Mixed Reality Educational Intervention
Behavioral: Traditional Breastfeeding Counseling — This intervention involves standard prenatal breastfeeding education provided by trained healthcare professionals. Participants receive verbal and visual explanations of breastfeeding techniques, benefits, and solutions to common challenges. Delivered in a single session during the third trimester of pregnancy, the session lasts approximately 60 minutes and represents the current standard of care in breastfeeding education.
  Arms: Traditional Breastfeeding Counseling

SUMMARY:
The goal of this randomized controlled trial is to evaluate whether a mixed reality-based educational strategy improves breastfeeding satisfaction and self-efficacy in pregnant women compared to traditional counseling. The study will involve women in their third trimester of pregnancy who are attending prenatal care in Sopó, Colombia.

The main questions it aims to answer are:

1. Does the mixed reality strategy increase maternal satisfaction with breastfeeding as measured by the Maternal Breastfeeding Evaluation Scale (MBFES)?
2. Does the mixed reality strategy enhance breastfeeding self-efficacy as measured by the Breastfeeding Self-Efficacy Scale-Short Form (BSES-SF)? Researchers will compare the mixed reality intervention to traditional counseling to see if it leads to higher satisfaction, self-efficacy, and adherence to exclusive breastfeeding during the first week of life.

Participants will: Receive either traditional counseling or the mixed reality educational intervention.

Complete self-reported surveys on breastfeeding satisfaction and self-efficacy at one week and one month postpartum.

Participate in follow-up calls to report breastfeeding practices, specifically adherence to exclusive breastfeeding during the first week postpartum.

This study aims to provide new insights into using innovative educational strategies to improve breastfeeding outcomes.

DETAILED DESCRIPTION:
This study is a randomized controlled trial designed to assess the impact of a mixed reality-based educational intervention on breastfeeding satisfaction and self-efficacy in pregnant women during their third trimester. The research will be conducted in Sopó, Colombia, where breastfeeding rates remain below recommended levels. The study aims to address key barriers, including maternal uncertainty and lack of confidence, which often hinder exclusive breastfeeding practices.

Participants will be randomly assigned to one of two groups:

Mixed Reality Intervention Group: This group will receive the traditional breastfeeding counseling offered during prenatal classes, supplemented by an innovative mixed reality educational strategy. This technology blends real-world scenarios with virtual elements, providing participants with a simulated breastfeeding experience. The intervention includes the use of mixed reality goggles, realistic breastfeeding mannequins, and immersive audio-visual tools to enhance learning and build confidence.

Traditional Counseling Group: This group will receive standard breastfeeding counseling as part of their routine prenatal care.

The primary outcomes of the study include:

Breastfeeding Satisfaction: Assessed using the Maternal Breastfeeding Evaluation Scale (MBFES), which evaluates maternal enjoyment, satisfaction with breastfeeding, and perceptions of the baby's growth and lifestyle adjustments.

Breastfeeding Self-Efficacy: Measured using the Breastfeeding Self-Efficacy Scale-Short Form (BSES-SF), focusing on maternal confidence, intention, and perceived capability to breastfeed successfully.

The secondary outcome will evaluate the percentage of newborns exclusively breastfed during the first week of life, measured through self-reported data collected via follow-up phone calls.

The study seeks to leverage the advantages of mixed reality technology to provide a practical, immersive, and emotionally engaging learning experience. It is anticipated that this approach will better prepare mothers for the challenges of breastfeeding, increase their confidence, and ultimately improve adherence to exclusive breastfeeding practices.

By comparing these two approaches, the trial aims to generate evidence that could inform future educational strategies, both locally and globally, for promoting breastfeeding and improving maternal and infant health outcomes.

ELIGIBILITY:
Inclusion Criteria:

Pregnant women in their third trimester enrolled in the prenatal care program. Aged 18 years or older, hemodynamically stable, conscious, and oriented.

Exclusion Criteria:

Pregnant or postpartum women and newborns with contraindications for breastfeeding (e.g., HIV positive, HTLV 1 or 2 positive, or undergoing chemotherapy for cancer).

Pregnant or postpartum women with intellectual or sensory disabilities. Newborns with congenital, anatomical malformations, or conditions that affect breastfeeding.

Admission of the mother or newborn to the neonatal intensive care unit (NICU).

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Self-identified females who are pregnant and meet the inclusion criteria are eligible to participate in this study.
Enrollment: 68 (Actual)
Dates: Start 2024-06-01 (Actual); Primary Completion 2024-12-01 (Actual); Study Completion 2025-01-10 (Actual)

PRIMARY OUTCOMES:
Score on Maternal Breastfeeding Evaluation Scale (MBFES) | From enrollment during the third trimester to the end of the first week postpartum
  Maternal Breastfeeding Evaluation Scale (MBFES): This scale includes 30 items assessing maternal enjoyment, satisfaction, infant growth, and maternal lifestyle. Responses are scored on a scale from 1 (strongly disagree) to 5 (strongly agree), with reverse scoring for negatively worded items. Total scores range from 30 to 150, with higher scores indicating greater breastfeeding satisfaction.
Breastfeeding Self-Efficacy Scale - Short Form (BSES-SF) | From enrollment during the third trimester to the end of the first week postpartum
  Breastfeeding Self-Efficacy Scale - Short Form (BSES-SF): This scale consists of 14 items evaluating maternal confidence, effort, thought patterns, and physical and psychological well-being. Responses range from 1 (never) to 5 (always), with total scores ranging from 14 to 70. Higher scores indicate greater self-efficacy in breastfeeding.

SECONDARY OUTCOMES:
Percentage of Neonates Exclusively Breastfed at Discharge and During the First Week of Life | From enrollment during the third trimester to the end of the first week postpartum.
  The secondary outcome is the percentage of neonates exclusively breastfed during two specific time points:
  At Discharge from Rooming-In:
  Mothers will report the type of feeding their newborns received during the hospital stay, focusing on exclusive breastfeeding without formula or other supplements.
  During the First Week of Life:
  A follow-up phone call will collect self-reported data on feeding practices during the first week postpartum, identifying whether the neonate was exclusively breastfed or received other feedings (e.g., formula or water).
  Exclusive breastfeeding is defined according to WHO guidelines, where the infant receives only breast milk, with no other liquids or solids except for oral rehydration solutions or medicines. The data will be analyzed to calculate the proportion of neonates exclusively breastfed at these two critical points.

CONTACTS AND LOCATIONS:
Overall Officials: Sergio Agudelo-Pérez, PhD. Assitent Proffesor, Principal Investigator — Universidad de la Sabana
Locations (1):
- Hospital de Sopo, Sopó, Cundinamarca, Colombia

REFERENCES:
- [Background] Tseng JF, Chen SR, Au HK, Chipojola R, Lee GT, Lee PH, Shyu ML, Kuo SY. Effectiveness of an integrated breastfeeding education program to improve self-efficacy and exclusive breastfeeding rate: A single-blind, randomised controlled study. Int J Nurs Stud. 2020 Nov;111:103770. doi: 10.1016/j.ijnurstu.2020.103770. Epub 2020 Sep 3. PMID 32961461
- [Derived] Montoya-Moncada A, Cuero-Rios L, Rodriguez-Morales F, Perdigon M, Agudelo-Perez S. Exploring the role of mixed reality education in maternal self efficacy and satisfaction with breastfeeding. Sci Rep. 2025 Aug 5;15(1):28484. doi: 10.1038/s41598-025-14319-y. PMID 40764648